CLINICAL TRIAL: NCT02999776
Title: An Observer Partially-blinded, Lesion-randomized, Intra-patient Controlled, 3-arm, Phase I Study to Assess Safety and Efficacy of Laser-assisted Topical Etanercept Administration in Patients With Mild to Moderate Plaque Psoriasis
Brief Title: Laser-assisted Topical Administration of Etanercept (Enbrel®) in Patients With Mild to Moderate Plaque-type Psoriasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pantec Biosolutions AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TopPso-2015
Record Dates: First submitted 2016-11-28; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Psoriatic Plaque
Keywords: Plaques Psoriasis; Topical; Laser microporation
MeSH Terms: interventions — betamethasone dipropionate, calcipotriol drug combination; Etanercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of care (Active Comparator): Daily self-administration of 1 to 5g Daivobet (Calcipotriol 50ug/g +Betamethasone, 0,5mg/g Gel) ointment, which is applied topically once per day for 8 weeks on one pre-selected randomized plaque.
  Interventions: Drug: Standard of care-daily administration of Daivobet
- Laser plus etanercept (Experimental): Immediately following microporation of a 5 cm² area of the designated plaque with the P.L.E.A.S.E.® Professional laser, 0.0625 ml of Etanercept (50 mg/ml) solution for injection in pre-filled syringes will be applied to the microporated surface of the lesion. The treated area will then be covered with OpSiteTM Flexigrid Transparent Dressing for 4 hours. This treatment procedure will be repeated twice weekly for 8 weeks.
  Interventions: Drug: Laser microporation + topical application of Etanercept
- Laser alone (Active Comparator): The Er:YAG laser induced microporation of 5 cm2 of a plaque surface, followed by application of an OpSiteTM Flexigrid Transparent Dressing for 4 hours. This treatment will also be repeated twice weekly for 8 weeks.
  Interventions: Device: Laser microporation alone

INTERVENTIONS:
Device: Laser microporation alone — The Er:YAG laser induced microporation of 5 cm2 of a plaque surface, followed by application of an OpSiteTM Flexigrid Transparent Dressing for 4 hours. This treatment will also be repeated twice weekly for 8 weeks.
  Other Names: P.L.E.A.S.E.
  Arms: Laser alone
Drug: Standard of care-daily administration of Daivobet — The other control treatment is Daivobet®, which is applied topically daily for 8 weeks on one pre-selected randomized plaque.
  Other Names: Daivobet
  Arms: Standard of care
Drug: Laser microporation + topical application of Etanercept — Immediately following microporation of a 5 cm² area of the designated plaque with the P.L.E.A.S.E.® Professional laser, 0.0625 ml of Etanercept (50 mg/ml) solution for injection in pre-filled syringes will be applied to the microporated surface of the lesion. The treated area will then be covered with OpSiteTM Flexigrid Transparent Dressing for 4 hours. This treatment procedure will be repeated twice weekly for 8 weeks.
  Other Names: Etanercept
  Arms: Laser plus etanercept

SUMMARY:
The purpose of this study is to assess the feasibility and safety of topical administration of etanercept via AFL micropores to psoriatic plaques in patients with mild to moderate plaque-type psoriasis.

While a wide variety of therapeutic innovations to treat moderate-to-severe psoriasis (accounting for around 30% of the cases) become available each year, there are few innovations for topical therapies to treat mild/localized psoriasis (accounting for around 70% of the cases). Given that only about half of the patients respond adequately to the current standard of care, the topical application of a fixed combination of calcipotriole and betamethasone, there is a medical need for better topical therapies.

Etanercept has been used successfully to treat moderate-to-severe plaque-type psoriasis in children and adults for more than a decade. Its standard route of application is through subcutaneous injections. Different dosing regimens have been used: 1 x 50 mg or 2 x 50 mg per week as well as 1 x 25 mg or 2 x 25 mg per week. Under these regimens, etanercept has a well-established favorable long-term safety record, with injection site reactions (pain, swelling) the most frequently reported side effects. However, rare but serious side effects such as serious opportunistic infections resulting from immune system inhibition common to anti-TNF agents limit its systemic use to these patients. For this reason, a localized topical alternative route of administration would be desirable. However, the large molecular size and chemical nature of etanercept prevent it from crossing the epidermal barrier. A CE certified ablative fractional laser (AFL) device with Er:YAG source will be used to create micropores in plaques to allow local delivery of etanercept directly into psoriatic plaques.

DETAILED DESCRIPTION:
Monocentric, observer partially-blinded Phase I study.

In this study, three similar plaques on each patient will be prospectively identified by the blinded observer and then randomized by an unblinded investigator by using the eCRF to one of the three study treatments:

1. Standard of care (daily administration of Daivobet® by the patient),
2. Ablative fractional laser microporation + topical application of etanercept
3. Ablative fractional laser microporation alone.

Over the treatment period of 8 weeks, patients will return to the clinic twice weekly for assessment of the three study plaques by the blinded observer, followed by administration of the treatment of plaques assigned to AFL microporation with or without etanercept. Patients will treat the remaining plaque with Daivobet® themselves on a daily basis.

Although no incompatibilities of AFL and etanercept are anticipated, because this is the first time etanercept is administered topically via AFL micropores and using a AFL microporation device, the study will be conducted in two stages: a Safety Stage consisting of the first five patients and the Study Stage with thirty patients.

In the Safety Stage of the study, three different plaques of the first 5 patients will be randomized and administered the respective treatments only once. Enrollment will be suspended after the 5th patient has been enrolled to permit the data monitoring committee (DMC) to review of the initial safety data from these first 5 patients to reassess risk. Based on this review, the DMC will make one of three recommendations:

1. to continue the study as planned,
2. to continue the study with adjustments to study procedures, such as changes to laser parameters, frequency of treatments or concentration of etanercept or,
3. in the event of extreme safety concerns, to terminate the study.

If option 1 is recommended, the study will resume with the Study Stage (Stage 2), in which the initial 5 patients will once again begin treatment, with their plaques receiving the same treatments to which they were previously randomized. Their treatment will continue for 8 weeks. Enrollment will also resume and continue until an additional 25 patients have been enrolled. If the DMC recommends option 2, treatment and enrollment will resume as just described after an adapted protocol has been submitted to and approved by the relevant authorities. If the DMC recommends option 3, then the study will terminate.

The Study Stage will consist of 2 periods: screening period (up to 2 weeks prior to baseline assessments and randomization) and treatment period (for the first 5 patients: initially 1 set of treatments, followed by suspension of treatment until after DMC review, then 8 weeks of treatment; for the remaining 25 patients: 8 weeks of treatment depending on plaque randomization, either daily Daivobet® or biweekly AFL with or without etanercept).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study related activity is performed.
2. Men or women, non-pregnant and non-lactating, at least 18 years of age at time of screening
3. Chronic mild to moderate plaque-type psoriasis diagnosed at least 6 months prior to baseline. Chronic mild to moderate plaque-type psoriasis as defined at screening by:

   * BSA affected by plaque-type psoriasis of less than 10%
4. Eligible for topical therapy according to current psoriasis treatment guidelines (12).

Exclusion Criteria:

1. Forms of psoriasis other than mild to moderate plaque-type (e.g., pustular, erythrodermic and guttate psoriasis)
2. Hyperpigmentation, e.g. birth marks, freckles, scar tissue at the psoriasis plaque areas that are intended to be treated
3. Intertriginous plaques or plaques on the hands, feet, neck, face, elbows, knees, or on the scalp will not be eligible as plaques for treatment.
4. Plaques on eyelids, lips or mucous membranes, open wounds, moles or birth marks, areas at risk of developing post-inflammatory hypo- or hyperpigmentation due to high levels of UV radiation subsequent to treatment will not be eligible for treatment.
5. Drug-induced psoriasis (i.e., new onset or current exacerbation from e.g. beta-blockers, or lithium)
6. Ongoing use of prohibited psoriasis treatments (e.g., topical corticosteroids, UV-therapy). Washout periods detailed in the protocol have to be adhered to (see Table 5-2)
7. Ongoing use of other non-psoriasis prohibited treatments. Washout periods detailed in the protocol have to be adhered to (see Table 5-2). All other prior non-psoriasis concomitant treatments must be on a stable dose for at least four weeks before baseline
8. Use of any other investigational drugs within 30 days prior to screening (or within 5 half-lives or until the expected PD effect has returned to baseline, whichever is longer).
9. Requiring treatment with any biological medicinal product during the study other than the study medication.
10. Any contraindication to etanercept (Enbrel®) or calcipotriol/betamethasone (Daivobet®).
11. Previous (last 12 months) and current exposure biologics, such as etanercept, adalimumab.
12. Any contraindication to treatment with the P.L.E.A.S.E® device, including Fitzpatrick skin types V or VI.
13. Current treatment or need for treatment with any prohibited medications (listed under Section 5.9.6).
14. Any serious illness or uncontrolled medical condition, including but not limited to severe infections, significant hepatic or renal disease, uncontrolled hypertension (defined as blood pressure ≥160/95), congestive heart failure (NYHA class III or IV), or other severe, uncontrolled cardiac disease.
15. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (cut-off as defined by laboratory)
16. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they agree to use highly effective methods of contraception (defined in Section 6.5.7) during the study and for 12 months after stopping treatment. Women are considered not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
17. Active ongoing inflammatory diseases other than psoriasis that might confound the evaluation of the benefit of treatment with etanercept
18. Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the patient and/or places the patient at unacceptable risk for receiving an immunomodulatory therapy
19. History of clinically significant liver disease or liver injury as indicated by abnormal liver function tests. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase may not exceed 2.5 x upper limit of normal at screening.
20. Pre-existing or recent-onset central or peripheral nervous system demyelinating disorders according to investigator's discretion and where necessary taking into account a neurological assessment; patients who are considered to have an increased risk of developing a demyelinating disease
21. Significant cardiovascular problems, including but not limited to the following: uncontrolled hypertension (blood pressure ≥160 systolic/95 diastolic mmHg), congestive heart failure with known decreased left ventricular ejection fraction
22. Patients with a serum creatinine level exceeding 176.8 μmol/L (2.0 mg/dL)
23. Any of the following laboratory values at screening: total WBC count <3,500/μL, or neutrophils <2,000/μL or platelets <125,000/μL or hemoglobin <10.0 g/dL
24. Positive serology to hepatitis C infection (i.e. positive antibody against Hepatitis C virus) or hepatitis B infection (i.e. positive hepatitis B surface antigen [HBsAg]).
25. Severely immunocompromised state, including but not limited to Felty's syndrome and known human immunodeficiency virus (HIV) infection
26. Active tuberculosis. If a QuantiFERON®- Tuberculosis (TB) Gold test at screening is positive, further work-up, according to local guidelines/practices needs to be performed to conclusively establish that that the patient has no evidence of active tuberculosis.
27. History of serious recurrent, chronic infectious disease (excluding fungal infections of the nail beds) or active systemic infections during the last two weeks (exception: common cold) prior to baseline and any infections that reoccur on a regular basis; patients with a history or evidence of opportunistic infections including specific pathogens such as listeria, legionella and parasitic infections. Investigator discretion should be used regarding patients who have traveled or resided in areas of endemic mycoses, such as histoplasmosis, coccidioidomycosis or blastomycosis and for patients with underlying conditions that may predispose them to infection, such as advanced or poorly controlled diabetes
28. Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C at screening or baseline
29. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system (except for basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 3 months, and except for carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed)
30. Current severe progressive or uncontrolled disease which in the judgment of the clinical investigator renders the patient unsuitable for the trial
31. Inability or unwillingness to undergo repeated venipuncture (poor tolerability or lack of access to veins)
32. Blood donation or blood loss of >400 ml in the 8 weeks prior to randomization.
33. History of hypersensitivity to any recombinant protein drugs or any of the excipients used in Enbrel® (see list of excipients in Table 5-1)
34. Patients who are allergic to rubber or latex (the needle cover on the prefilled syringes for Enbrel® contain dry natural rubber)
35. Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol
36. History or evidence of ongoing alcohol or drug abuse, within the last six months before baseline
37. Plans for administration of live vaccines during the study period or live vaccination within 6 weeks prior to baseline
38. Patients not willing to limit UV light exposure (e.g., sunbathing and/or the use of tanning devices) during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Administration site reactions (ASR) | 8 weeks
  The investigator or qualified designee will assess ASRs such as itching, redness, swelling, pain, or ulceration at time points as indicated in Table 6-1. Whenever possible, the same evaluator should perform this assessment at all visits and document the result in the eCRF. An ASR that fulfills the criteria of an SAE should be documented and reported as such.

SECONDARY OUTCOMES:
Target Plaque Severity Score (TPSS) | 8 weeks
  The blinded observer will perform the TPSS assessment at baseline (Visit 2) and at treatment visits 9 and 18. Whenever possible, the same evaluator should perform this assessment at all visits. For TPSS assessment, the target plaques will be evaluated separately for induration, scaling and erythema using a 5-point severity scale.

CONTACTS AND LOCATIONS:
Overall Officials: Wolf-Henning Boehncke, Prof., Principal Investigator — HUG
Locations (1):
- University Hospital Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No